CLINICAL TRIAL: NCT03984266
Title: The Pre-clinical Study of Genomic Sequencing for Birth Defects in Newborns
Brief Title: The Pilot Study of High-throughput Sequencing in Neonatal Birth Defects
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Collaborators: Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); Maternal and Child Health Hospital of Hubei Province (Other); The First Hospital of Jilin University (Other); Xuzhou Maternity and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Xia Yunqiu, Research assitant, Children's Hospital of Chongqing Medical University
Other Study IDs: CHCMU-CCMM-01
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Birth Defect; Newborn; Fit; Genetic Diseases; Multiple Malformation; Congenital Malformation
MeSH Terms: conditions — Congenital Abnormalities; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: NGS panel — A next-generation-sequencing panel, which contains a group of genes that specifically cause disease, for mutational analysis in newborns.

SUMMARY:
In China, birth defects can reach as high as 5.6%, about 900,000 new cases of birth defects are added each year, making it the second cause of death for infants, with a total death rate of 19.1%. At present, China implements the three-level prevention and control system for birth defects, which is performed before marriage, before birth, and during the neonatal period. Newborn screening is the last line of defense against birth defects. Early screening diagnosis and timely intervention are extremely important, especially for diseases which can be preventive and treatable. This study aims to evaluate the clinical application of high-throughput targeting sequencing in newborns, and investigate whether this new technology can significantly shorten the time of examination, improve the diagnosis rate, guide the intervention treatments and promote prognosis for these disease.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates in one of the study hospitals
2. Abnormal laboratory testing or abnormal response to standard therapy suggestive of a genetic disease

Exclusion Criteria:

1. Any infant whose genome has been shown to have large chromosomal aberration (Trisomy 13, 18, 21 or other)
2. Any infant in which clinical considerations preclude drawing 1.0 ml of peripheral blood
3. Parents refuse consent

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates in one of the study hospitals
Sampling Method: Non-Probability Sample
Enrollment: 3423 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | At corrected age of 18 months
  Incidence of death
Disability Rate | At corrected age of 18 months
  Incidence of disability. Disability defined as a physical or mental handicap, especially one that prevents a person from living a full, normal life or from holding a gainful job.
Allele Frequency | In 120 days after receipt of all the patients' sequencing data
  Allele frequency, or gene frequency, is the relative frequency of an allele (variant of a gene) at a particular locus in the population the investigators studied, expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zou, Ph.D, Study Chair — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Yes